CLINICAL TRIAL: NCT03532997
Title: Developing and Testing a Web-based Tool to Engage Advanced Cancer Patients in Palliative Care (ēlos)
Brief Title: Extra Layer Of Support
Acronym: ELOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00089227
Record Dates: First submitted 2018-05-10; First posted 2018-05-22 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Advanced Cancer; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The investigators aim to introduce patients with advanced cancer to supportive care resources, including specialty palliative care, through a novel app called "ELOS" (stands for "extra layer of support) in a prospective cohort study. The investigators will compare participant acceptance of this new electronic tool to industry standards and follow ultimate referrals to outpatient palliative care compared to historical, matched controls.
  Interventions: Other: ELOS

INTERVENTIONS:
Other: ELOS — The investigators aim to introduce patients with advanced cancer to supportive care resources, including specialty palliative care, through a novel web-based application called "ELOS" (stands for "extra layer of support) in a prospective cohort study.

SUMMARY:
The investigators aim to introduce patients with advanced cancer to supportive care resources, including specialty palliative care, through a novel app called "ELOS" (stands for "extra layer of support) in a prospective cohort study. The investigators will compare participant acceptance of this new electronic tool to industry standards and follow ultimate referrals to outpatient palliative care compared to historical, matched controls.

DETAILED DESCRIPTION:
The investigators will conduct a prospective cohort study to investigate usability of implementing Ēlos across 50 advanced cancer patients within the Duke Cancer Institute and University of North Carolina - Chapel Hill Cancer Center. The investigators will obtain a Data Transfer Agreement prior to enrollment at the University of North Carolina. Usability testing evaluates a technology system's capacity for practical implementation in the field including logistical, social, financial, regulatory, and time considerations. The Usability test will also build foundational data needed to design a future, multi-site controlled trial evaluating the efficacy of Ēlos alongside exploring real-world implementation issues to address prior to undertaking the larger trial.

To conduct the study, the investigators will consecutively approach two populations: adult advanced cancer patients (defined as any Stage IV solid tumor malignancy, or Stage III pancreas or lung cancer) in the GI, GU, and Thoracic Cancer Clinics with a diagnosis made in the preceding eight weeks. The investigators will primarily evaluate usability through evaluating subject-reported perceived usefulness. .

The investigators will also measure change in patient self-efficacy and change knowledge of palliative care scores alongside obtaining baseline data on palliative care referral rates.

To evaluate perceived usefulness, the investigators will use the Perceived Usefulness Scale and Ease of Use subscales of the System Usability Scale, common tools used in health technology evaluations30 and a single item "I feel prepared for the palliative care visit".

Lastly, the investigators will measure subsequent referrals to palliative care, comparing the Ēlos cohort with a non-intervention cohort. the investigators will compare three cohorts: 1). Ēlos intervention cohort; 2). An age-, disease-, and stage-matched cohort of usual care patients during the same time period as the intervention; and 3). A similarly-matched cohort who received usual oncology care six months prior to the study. The latter control cohort evaluates palliative care referral practices prior to any intervention taking place to reduce contamination. The investigators will use these preliminary data on referral rates to determine the effect sizes needed to calculate the sample sizes for an Alliance CCDR protocol for a NCORP trial.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* capacity to give consent
* has received a diagnosis of Stage IV solid tumor malignancy or Stage III pancreas or lung cancer within the 8 weeks prior to consent
* ability to speak and understand English
* has access to a computer and the internet

Exclusion Criteria:

* Not Age 18 or older
* Does not have capacity to give consent
* Has not received a diagnosis of Stage IV solid tumor malignancy or Stage III pancreas or lung cancer within the 8 weeks prior to consent
* Does not have the ability to speak and understand English
* Does not have access to a computer and the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Usability as measured by the System Usability Scale | Up to one hour
  The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking.
Validity as measured by the symptom assessment module | Up to one hour
Change in Palliative Care referral | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center - Cancer Prevention, Detection and Control, Durham, North Carolina, United States